CLINICAL TRIAL: NCT06279182
Title: The Impact of Barre Stretching on Self-Reported Stress and Pain Levels Among Entry-Level Dental Hygiene Students
Brief Title: Impact of Barre Stretching Among Dental Hygiene Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Idaho State University (Other)
Responsible Party: Principal Investigator, Vanessa Whiley, Principle Investigator, Idaho State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-FY2024-106
Record Dates: First submitted 2024-01-29; First posted 2024-02-26 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Musculoskeletal Disorders; Stress Management; Perceived Stress; Reported Stress; Perceived Pain; Reported Pain
Keywords: dental hygiene students; ergonomics; prevention; stretching; barre
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: The experimental group will receive the Barre stretching intervention. The control group will not receive any intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Barre Stretching Intervention (Experimental): 15 minute Barre stretching video two times a week for 6 weeks.
  Interventions: Behavioral: Barre Stretching Intervention
- Control Group: No Intervention (No Intervention): Participants do not participate in the Barre stretching intervention.

INTERVENTIONS:
Behavioral: Barre Stretching Intervention — The Barre stretching intervention will consist of a 15-minute recorded video session with static and isometric movements focused on the hands, wrists, shoulders, and neck combined with breathing exercises throughout each movement. A 15-minute Barre stretching video will be selected for this study because static and isometric stretching should be held for 10-15 seconds per movement and repeated 2-3 times for increasing blood flow and circulation which can improve heart rate variability (HRV), increase muscle suppleness in preparation for muscle activation through patient care, and reduce stress levels through regulation of the rate, depth, and pattern of breathing. The duration of 15-minutes provided the participants with adequate time to complete each stretching movement for a total of 45 seconds with 15 seconds rest between movements. There will be fifteen targeted stretching movements focused on the hands, wrists, shoulders, and neck region.
  Arms: Barre Stretching Intervention

SUMMARY:
The healthcare profession of dental hygiene can be a highly stressful academic path and occupation. Physical stressors can quickly lead to postural disturbances and musculoskeletal disorders (MSDs) due to instrument grasping while under muscle tension, working with vibrating instruments, and performing repetitive micromovements. Chronic, high stress levels have the potential to lead to burnout, fatigue, and other health problems, which can impact a student's ability to perform well in their clinical rotations and didactic studies and may translate into their workforce experiences after graduation.

The purpose of this study is to determine whether a relationship exists between Barre stretching and reported stress and pain levels among entry-level dental hygiene students.

This study will be a 6-week experimental randomized control trial (RCT) where participants will be assigned to a 15-minute Barre stretching and breathing video two times a week for the experimental group or control group. The continuous dependent variables in this study will be the reported stress levels and reported pain levels of the entry-level dental hygiene students. The independent variable will be the Barre stretching intervention. The participants will include students at two universities enrolled in an entry-level dental hygiene program as first-year students.

Baseline data collection for each participant will be obtained, and the study will be analyzed using descriptive statistics, a paired t-test and independent t-test. The statistical significance level will be set at p=0.05.

DETAILED DESCRIPTION:
Due to the unknown relationship between Barre stretching and dental hygiene students' reported stress and pain levels, the purpose of this research study is to determine whether relationships exist between implementing a Barre stretching and breathing routine to reduce this demographics' reported stress and pain levels. As technological advancements and patient centered care continue to drive the dental profession, hygienists continue to face challenges related to providing safe dental care for their patients and as practitioners while managing stress. This methodology chapter discusses the study's design, research sample, setting, data collection, statistical analysis, and limitations.

Overview of Study Research Questions. The following research questions guided the conduct of this study.

1. What are the self-reported stress levels among first-year dental hygiene students regarding job-related musculoskeletal training before and after participation in a 6-week regimented Barre stretching program?
2. What are the self-reported pain levels among first-year dental hygiene students regarding job-related musculoskeletal training before and after participation in a 6-week regimented Barre stretching program?

Hypotheses. The two-hypothesis related to this study are:

H1: Entry-level dental hygiene students who participate in a 6-week Barre stretching intervention will have statistically significant reduced levels of self-reported stress compared to those entry-level dental hygiene students who do not participate in the Barre intervention.

Ho: There is no significant difference in self-reported stress levels of entry-level dental hygiene students after participating in a 6-week Barre stretching intervention as compared to entry-level dental hygiene students who do not participate in the Barre intervention.

H1: Entry-level dental hygiene students who participate in a 6-week Barre stretching intervention will have statistically significant reduced levels of self-reported stress compared to those entry-level dental hygiene students who do not participate in the Barre intervention.

Ho: There is no significant difference in self-reported pain of entry-level dental hygiene students after participating in a 6-week Barre stretching intervention as compared to entry-level dental hygiene students who do not participate in the Barre intervention.

Variables The continuous dependent variables in this study will be the self-reported stress and pain levels of the entry-level dental hygiene students. The categorical dependent variables will be the Perceived Stress Scale (PSS-10) and the Numerical Rating Pain Scale (NRPS-11). The independent variable will be the Barre stretching intervention.

Research Design This study will be an experimental randomized control trial (RCT). A randomized control trial is a prospective study where data is collected over time and participants are tracked to measure the effectiveness of a new treatment or intervention. A RCT was selected for this study to investigate the research questions to evaluate differences between the experimental and control groups, while reducing bias and establishing a cause-effect relationship between the intervention and the outcome. This experimental RCT will have a two-group pre-and post-test design. Baseline data collection for each participant will be obtained, and the study will be analyzed using descriptive statistics, a paired t-test and independent t-test. The statistical significance level will be set at p=0.05. The CONSORT checklist when reporting a pilot or feasibility study will be used as a guide for this study.

Research Context The participants will include Idaho State University students enrolled in an entry-level dental hygiene program as first-year students. This institution will provide good prospects for a sample study of participants due to a highly competitive application process and baccalaureate degree completion.

Research Participants Sample Description. A convenience sample of students from Idaho State University's Department of Dental Hygiene baccalaureate program's first-year entry-level dental hygiene students will be invited to participate in the study. A convenience sample will be utilized to represent entry-level dental hygiene students who are new to the profession of dental hygiene and likely unaware of ergonomics and work-related musculoskeletal disorder risks, and potentially in a stressful time of their robust curriculum. Although convenience samples are non-probability sampling methods, they are widely used in clinical educational research and the most applicable for the purpose of this study based on subject availability and accessibility of entry-level dental hygiene students.

The participants for this research study were recruited after email contact was established through their program directors and lead clinical instructors at Idaho State University. An introduction of the study outlining its purpose and student involvement was presented, including an informed consent, followed by a health history pre-screening form, if qualified. The participating entry-level dental hygiene student's pre-screening medical histories will be reviewed to identify pre-existing conditions that might disqualify students from participating in the study.

Inclusion criteria. Participants of this convenience sample will be entry-level dental hygiene students (aged 18 or over) without any significant health limitations that will prevent the student from participating in Barre stretching movements.

Exclusion criteria. Entry-level dental hygiene student individuals who are under the age of 18 and with significant health limitations that will prevent them from participating in Barre stretching movements, will not be included in the study. Significant health conditions will include unstable joints or recent joint replacements and/or history of back/spinal injuries. Significant health conditions deeming participants exempt from participation will include unstable joints or recent joint replacements, and/or history of back/spinal injuries.

Human Subjects Protection. The proposal will be submitted to the Human Subjects Committee at Idaho State University for approval. Once approved by the Human Subjects Committee at Idaho State University, the study will be registered for a clinical trial number through clinicaltrials.gov. Additionally, after approval is given, a pre-intervention medical history will be completed by participants to identify if participants will meet the study inclusion criteria. Eligible participants' consent will be obtained via written consent form.

Data Collection. Qualifying participants will be asked to complete the Perceived Stress Scale (PSS-10) to establish self-reported stress levels and the Numerical Rating Pain Scale (NRPS-11) to establish self-reported pain levels prior to participating in either the control group or the intervention group. Participants will be divided into an even distribution of participants in either the intervention or control group. The post-test will be administered to the participants through published content through their universities individual learning management systems, Moodle and Canvas, respectively.

Instruments. The instrument to measure pain levels will be the Numerical Rating Pain Scale (NRPS-11), a self-reported pain survey, and the Perceived Stress Scale (PSS-10), a self-reported stress survey. Written permission was stated and given for use of the NRPS-11 and PSS-10 scales for educational and clinical research. Self-reported PSS-10 and NRPS-11 questionnaires will be provided to the students at the beginning of their Fall semester term, through their learning management systems to complete electronically, Idaho State University utilizes the platform called Moodle. The 6-week Barre stretching intervention instructional video will be published for students to access their individual learning management systems and will be completed two times a week (Monday and Thursday).

Procedure and Protocols. The participants will be assigned into a control group or experimental group through a computer-generated random assignment generator, Research Randomizer. The experimental group will receive the Barre stretching intervention. Since the Barre stretching video session will be online, the students will be instructed to complete it in a quiet, comfortable setting. The trial's intention is to create a relaxed session environment which disrupted the student's learning environment as little as possible, without affecting the outcome of the study. The Barre stretching intervention will consist of a 15-minute recorded video session with static and isometric movements focused on the hands, wrists, shoulders, and neck combined with breathing exercises throughout each movement. A 15-minute Barre stretching video will be selected for this study because static and isometric stretching should be held for 10-15 seconds per movement and repeated 2-3 times for increasing blood flow and circulation which can improve heart rate variability (HRV), increase muscle suppleness in preparation for muscle activation through patient care, and reduce stress levels through regulation of the rate, depth, and pattern of breathing. The duration of 15-minutes provided the participants with adequate time to complete each stretching movement for a total of 45 seconds with 15 seconds rest between movements. There will be fifteen targeted stretching movements focused on the hands, wrists, shoulders, and neck region.

Reliability and Validity. The PSS-10 perceived stress scale was selected for this study due to demonstrated adequate internal consistency (Cronbach's Alpha = .87), hypothesis testing [HEALTH (r = -.37); MENT (r = -.32); PHYS (= -.24)], and test-retest reliability (.86). The PSS-10 scale is a stress assessment instrument that consists of ten Likert-scale questions intended to measure current life situations represented as unpredictable and/or uncontrollable. The NPRS-11 is a pain assessment instrument that consists of an 11-point Likert scale used to measure self-reported pain among adult populations. The participant will select a whole number (0-10) that best reflects the intensity of their reported pain, with 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-9 = severe pain, and 10 = extreme pain/worst pain possible. The NPRS-11 was selected for this study due to demonstrated high test-retest reliability (r = 0.82) and correlation validity of the NPRS and VAS (r = 0.941).

Limitations. There may be limitations to this study, which include a smaller sample size (n=11), which limits the capacity of the statistical analysis. Another limitation is the selection of a convenience sample of entry-level dental hygiene students.

This RCT study collected two forms of data amongst entry-level dental hygiene students: self-reported stress levels (PSS-10) and self-reported pain levels (NRPS-11). The findings of this study addressed the research objective listed by the National Dental Hygiene Research Agenda related to occupational health, focused on "career satisfaction and longevity research assessing the dissemination and translation into practice methods that reduce the harmful effects of occupational stressors on practitioners." This RCT will address Healthy People 2030 objectives centered around improving public health issues using science-based objectives to increase the proportion of adults who engage in physical activity for substantial health benefits (PA-02, PA-03, PA-04, and PA-05). The results and discussion manuscript will be reported in the form of a manuscript to be submitted for publication in the International Journal of Dental Hygiene. The remaining sections of the thesis reflect the manuscript specifications outlined in the author guidelines located at https:www.adha.org/journal-of-dental-hygiene/.

ELIGIBILITY:
Inclusion Criteria:

* Participants of this convenience sample will be entry-level dental hygiene students (aged 18 or over) without any significant health limitations that will prevent the student from participating in Barre stretching movements.

Exclusion Criteria:

* Entry-level dental hygiene student individuals who are under the age of 18 and with significant health limitations that will prevent them from participating in Barre stretching movements, will not be included in the study. Significant health conditions will include unstable joints or recent joint replacements and/or history of back/spinal injuries. Significant health conditions deeming participants exempt from participation will include unstable joints or recent joint replacements, and/or history of back/spinal injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Self-Reported Stress (Perceived Stress Scale) | 6 weeks
  A change in the pre-to-post perceived stress test scores (likert scale 1-10: 1 being better, 10 being worst values).
Self-Reported Pain (Numerical Pain Rating Scale/Visual Analog Scale) | 6 weeks
  A change in the pre-to-post perceived pain test scores (likert scale 0-10: 0 being no pain, 10 being worst pain possible).

CONTACTS AND LOCATIONS:
Locations (1):
- Idaho State University, Pocatello, Idaho, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT06279182/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT06279182/ICF_001.pdf